CLINICAL TRIAL: NCT04192682
Title: Anlotinib Combined With Sintilimab as Second-line Treatment or Beyond in Patients With Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changzhou Cancer Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHSU2019011
Record Dates: First submitted 2019-04-22; First posted 2019-12-10 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Anlotinib; Sintilimab; Third-line Treatment or Beyond
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Combined With Sintilimab (Experimental): Anlotinib Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle, Combined With Sintilimab 200mg/time，21-day cycle。
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Anlotinib Day 1 to day 14 followed by 7 days off treatment in a 21-day cycle, Combined With Sintilimab 200mg/time，21-day cycle。
  Other Names: Sintilimab

SUMMARY:
Immunotherapy combined with anti-angiogenic therapy can achieve better results in patients with second-line and above small cell lung cancer

DETAILED DESCRIPTION:
Through this study, it was found that Anlotinib combined with Sintilimab has a better survival benefit. At the same time, genetic analysis and immunohistochemical methods have been used to predict the predictive value of targeted therapy combined with Sintilimab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should participate in the study voluntarily and sign informed consent;
2. Male or female aged over 18 years;
3. Histological documentation of small cell lung cancer
4. Advanced small cell lung cancer who failed first-line chemotherapy ,at least one measurable lesion (by RECIST1.1)
5. ECOG PS:0-2,.
6. Life expectancy of more than 3 months
7. The laboratory results at the screening point must meet the following requirements:

   (a) Blood routine: the absolute neutrophile count (ANC) shoud be more than 1.0 x 109/L, the platelet count (PLT) should be more than 100 x 109/L, the hemoglobin (HGB) should be more than 90g/L (no blood transfusion or erythropoietin dependence within 7 days);

   B) Liver function: total bilirubin (TBIL) should be less than or equal to 1.5 times of the upper limit of normal (ULN); avoid the subjects with liver metastasis, who had the levels of ALT and AST less than the 2.5 times of ULN; and the levels of ALT and AST in subjects with liver metastasis should less than the 5 times of ULN;

   C) Renal function: the level of serum creatinine (Cr) should less than 1.5 times of ULN or the clearance ratio of Cr should higher than 60 mL/min

   (Cockcroft-Gault formula) and the test results of urine routine showed the urine protein (UPRO) content should less than 2 + or should less than 1 g at the 24-hour urinary protein quantification;
8. For female subjects with reproductive age, the urine or serum pregnancy test should be negative within three days before receiving the first administration of the researched drug (the first cycle, first day). If the urine pregnatncy test is not enough to confirm the negative results, then the blood pregnancy test is required.
9. The compliance of the research programs is expected to be good.

Exclusion Criteria:

1. Patients who have been used anlotinib or Sintilimab;
2. Other malignant tumors (except clinically cured cervical carcinoma in situ, basal cell or squamous cell skin cancer and papillary thyroid cancer) that were concurrently diagnosed or have occurred within 5 years.
3. The patients who had received chemotherapy, radiotherapy or other experimental anticancer therapy within 4 weeks before treatment; those who had received local radiotherapy in the past could be included in this research, if the following conditions were meet: radiotherapy was performed more than 4 weeks before the beginning of this study (brain radiotherapy was performed more than 2 weeks), and the target lesions selected in this study were not in the radiotherapy area, or the target lesions were in the radiotherapy area, but the progress was confirmed.
4. Systematic systemic treatment with Chinese herbal medicine or immunomodulatory drugs (including thymosin, interferon and interleukin, except for local use of pleural effusion) was given within 2 weeks before the first administration.
5. Received live attenuated vaccine within 4 weeks before the first administration (or planned to receive live vaccine during the study period);

   Note: Inactivated (killed) virus vaccines for seasonal influenza are allowed within 4 weeks before the first administration, but live attenuated influenza vaccines are not allowed.
6. Patients had undergone large and medium-sized operations or unhealed surgical incisions, ulcers or fractures within 4 weeks before the first administration.
7. Patients who were undergoing any other forms of immunosuppressive therapy, not including local glucocorticoids or physiological dose of systemic glucocorticoids (<10 mg/day prednisone or equivalent doses of glucocorticoids) through nasal spray, inhalation or other routes, within 7 days before the first administration.
8. Patients had a history of non-infectious pneumonia requiring glucocorticoid therapy or currently have interstitial lung disease one year before the first administration.
9. Active autoimmune diseases requiring systemic treatment (e.g. using the disease-relieving drugs, corticosteroids or immunosuppressants) occurred within two years before the first administration. Allow the use of alternative therapies (such as thyroxine, insulin or physiological corticosteroids for adrenal or pituitary insufficiencies).
10. Patients with Asymptomatic central nervous metastasis; For patients who had stable symptoms (> 2 weeks) after treatment of brain metastases, they can participate in this study as long as they meet all the following criteria: there are measurable lesions outside the central nervous system; no metastases of the midbrain, pons, cerebellum, medulla oblongata or spinal cord; no history of intracranial hemorrhage in the past; stop the discontinuation of hormone therapy 7 days before the medication treatment;
11. Before the start of treatment, patients who had not been fully recovered from the toxicity and/or complications caused by any intervention (i.e., less than grade 1 or reaching the baseline, excluding fatigue or alopecia);
12. Patients who had the uncontrollable third interstitial effusion (e.g. pleural effusion/pericardial effusion).
13. Patients who had any unstable systemic disease: including but not limited to active infections, unstable angina pectoris, cerebrovascular accident or transient ischemic attack (within 6 months before screening), myocardial infarction (within 6 months before screening), congestive heart failure [New York Heart Association (NYHA) Classification >Class II], severe arrhythmias requiring medication treatment, liver, kidney or metabolic disease;
14. Patients who had received solid organ or blood system transplantation, except corneal transplantation.
15. A known history of human immunodeficiency virus (HIV) infection (i.e. positive HIV 1/2 antibody);
16. Active or current tuberculosis requiring medical intervention, including but not limited to tuberculosis;
17. Patients who had untreated active hepatitis B; Note: Hepatitis B patients could be included in this research if they meet the following criteria:
18. The hepatitis B virus (HBV) load must be less than 1000 copies/ml (200 IU/ml) before the first administration. Anti-HBV therapy should be taken throughout the study period to avoid viral reactivation. For subjects who had HBcAb (+), HBsAg (-), HBsAb (-), HBsAb (-) and HBV viral load (-), no prophylactic anti-HBV treatment is required, but virus reactivation needs to be closely monitored.
19. Subjects with active hepatitis c virus (HCV) infection (HCV antibody positive and HCV-RNA level higher than the detection limit);
20. Subjects who had severe allergic reactions (> grade 3) to the active ingredients and any excipients of Sindelimab, Anlotinib hydrochloride.
21. Pregnant or lactating women or women preparing for pregnancy or lactation during the study period;
22. For men or women at risk of conception, and they disagree with the application of effective contraception during the study period and within 90 days after the last administration.
23. Patients who had a history of alcoholism or drug abuse;
24. Other conditions that researchers considered not suitable for including in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | At least 1 year following the conclusion of immunotherapy
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Overall Survival | At least 1 year following the conclusion of immunotherapy
  Overall Survival is defined as the length of time from random assignment to death or to last contact.
Objective Response Rate | At least 1 year following the conclusion of immunotherapy
  Objective response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）

CONTACTS AND LOCATIONS:
Overall Officials: Tong Zhou, Principal Investigator — Changzhou Cancer Hospital of Soochow University
Locations (1):
- Changzhou Cancer Hospital of Soochow University, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No